CLINICAL TRIAL: NCT01128530
Title: A Randomized, Controlled, Double-Blind, Double Dummy, Multicenter Phase 2 Study of the Safety/Tolerability and Efficacy of JNJ-32729463 Compared With Linezolid (Zyvox) for the Treatment of Complicated Skin and Skin Structure Infection
Brief Title: Efficacy and Safety Study of JNJ-32729463 for Treating Complicated Skin and Skin Structure Infections Compared to Linezolid (Zyvox)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Furiex Pharmaceuticals, Inc (Industry)
Responsible Party: June Almenoff, MD, President/CMO, Furiex Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32729463CSI2001
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Complicated Skin and Skin Structure Infections
Keywords: cSSSI; complicated skin and skin structure infections; acute bacterial skin and skin structure infections; abscess; cellulitis; bacterial infections; anti-bacterial agents; anti-infective agents; skin diseases, infectious; skin diseases; wound infection
MeSH Terms: conditions — Abscess; Cellulitis; Bacterial Infections; Skin Diseases, Infectious; Skin Diseases; Wound Infection | interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-32729463 (Experimental): JNJ-32729463 250 mg tablet and matching linezolid placebo twice daily
  Interventions: Drug: JNJ-32729463; Drug: linezolid placebo
- linezolid (Active Comparator): linezolid 600 mg tablet and matching JNJ-32729463 placebo twice daily
  Interventions: Drug: linezolid; Drug: JNJ-32729463 placebo

INTERVENTIONS:
Drug: JNJ-32729463 — 250 mg tablet twice daily
  Arms: JNJ-32729463
Drug: linezolid — 600 mg tablet twice daily
  Other Names: Zyvox
  Arms: linezolid
Drug: JNJ-32729463 placebo — 1 placebo tablet twice daily
  Arms: linezolid
Drug: linezolid placebo — 1 placebo tablet, twice daily
  Arms: JNJ-32729463

SUMMARY:
The purpose of this study is to determine the clinical efficacy, safety, and tolerability of a 250 mg BID oral dose of JNJ-32729463 compared with linezolid in subjects with complicated skin and skin structure infections (cSSSIs).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a complicated skin and skin structure infection (cSSSI) including wound infection, deep cellulitis or severe abscess
* Women of childbearing potential must agree to use an acceptable form of contraception
* Infection site offers ability to obtain a microbiological specimen
* Received only 1 dose of any potentially effective systemic antibiotic within 24 hours of beginning study treatment

Exclusion Criteria:

* History of hypersensitivity or allergic reaction to quinolones or to linezolid
* Female and pregnant or breastfeeding or may be pregnant
* Chronic or underlying skin condition surrounding the area of infection that may complicate the assessment of response (e.g. atopic dermatitis, eczema, or psoriasis)
* Subject has infections with a high cure rate after surgical incision alone after aggressive local skin care
* Subject has infection(s) suspected to be caused by Gram-negative rods, anaerobic bacteria or unusual pathogens
* Subject has an infection that is expected to require other antifungal, antimycobacterial, or antibacterial agents in addition to study medication

Other protocol-specific eligibility criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cessation of spread or reduction in the size of the primary infection site lesion | 48-72 hours
Defervescence | 48 - 72 hours

SECONDARY OUTCOMES:
Severity of signs and symptoms of the primary infection site lesion | up to day 84-98 (late follow-up visit)
Clinical response rate - overall and for MRSA | Day 10 (TOC visit), Day 15-21 (SFU/EOT visit)
Microbiological response rate - overall and for MRSA | Day 15-21 (SFU/EOT visit)
Change in susceptibility testing of S. aureus | Day 15-21 (SFU/EOT visit)
  Changes in susceptibility testing of S. aureus isolates from the original infection site to linezolid and JNJ-32729463
Rate of recurrence and new infection in subjects with MRSA | Day 35-49 and Day 84-98
Defervescence | Day 4 (Visit 3)
Cessation of spread or reduction in the size of the primary infection site lesion | Day 4 (Visit 3)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Furiex Research Site, Anaheim, California
  - Furiex Research Site, Buena Park, California
  - Furiex Research Site, Chula Vista, California
  - Furiex Research Site, Fountain Valley, California
  - Furiex Research Site, La Mesa, California
  - Furiex Research Site, Long Beach, California
  - Furiex Research Site, Oceanside, California
  - Furiex Research Site, Santa Ana, California
  - Furiex Research Site, Fort Myers, Florida
  - Furiex Research Site, Kissimmee, Florida
  - Furiex Research Site, Saint Cloud, Florida
  - Furiex Research Site, Columbus, Georgia
  - Furiex Research Site, Savannah, Georgia
  - Furiex Research Site, Idaho Falls, Idaho
  - Furiex Research Site, Libertyville, Illinois
  - Furiex Research Site, Baton Rouge, Louisiana
  - Furiex Research Site, New Orleans, Louisiana
  - Furiex Research Site, Sulphur, Louisiana
  - Furiex Research Site, Detroit, Michigan
  - Furiex Research Site, Keego Harbor, Michigan
  - Furiex Research Site, Butte, Montana
  - Furiex Research Site, Toledo, Ohio
  - Furiex Research Site, Philadelphia, Pennsylvania
  - Furiex Research Site, Houston, Texas
  - Furiex Research Site, Sugar Land, Texas
  - Furiex Research Site, Webster, Texas